CLINICAL TRIAL: NCT01671670
Title: Phase III Study of Acupuncture for Patients With Functional Dyspepsia
Brief Title: Acupuncture for Patients With Function Dyspepsia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Collaborators: Hunan University of Traditional Chinese Medicine (Other); Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012CB518501-3; 2012CB518501 (Other Grant/Funding Number: The Chinese Ministry of science and technology)
Record Dates: First submitted 2012-08-21; First posted 2012-08-23 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Functional Dyspepsia; Postprandial Distress Syndrome
Keywords: Functional dyspepsia; postprandial distress syndrome
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acupuncture group (Experimental): use traditional acupuncture to treat functional dyspepsia
  Interventions: Other: acupuncture
- sham acupuncture group (Sham Comparator): use penetrating sham acupuncture to manage functional dyspepsia
  Interventions: Other: sham acupuncture

INTERVENTIONS:
Other: acupuncture — In this group, acupuncture is given according to traditional acupuncture theories.
  Other Names: use hwato acupuncture needles
  Arms: acupuncture group
Other: sham acupuncture — Sham acupuncture points will be used in this trial, with needle penetration.
  Other Names: verum acupuncture
  Arms: sham acupuncture group

SUMMARY:
Hypothesis: Acupuncture is efficacious and safe for patients with functional dyspepsia

Design:

* A single blind randomized controlled trial
* 200 participants will be included
* Two arms: acupuncture and sham acupuncture group

DETAILED DESCRIPTION:
Aim: to clarify the efficacy and safety of acupuncture for patients with functional dyspepsia Design: A single blind randomized controlled trial will be performed in Chengdu, Hunan and Chongqing province. Two hundred participants will be randomly assign to acupuncture and sham acupuncture group. Each participants will receive 20 sessions of acupuncture in 4 weeks, with a duration of 30 minutes in a session. The primary outcome is Patients' global assessments of efficacy in 16 weeks after inclusion. Secondary outcomes include validated Leeds Dyspepsia Questionnaire, Nepean dyspepsia index, etc.

ELIGIBILITY:
Inclusion Criteria:

* Consistent with the diagnostic criteria of functional dyspepsia.
* Age of a subject is older than 18 and is younger than 65.（including 18 and 65）
* Include postprandial distress syndrome.
* Did not take any gastroenteric dynamic drugs in the last 15 days, and did not take part in any clinical trial.
* Informed consent is signed by a subject or his lineal relation.

Exclusion Criteria:

* Patients with any contraindications of Itopride.
* Patients who are unconscious, psychotic.
* Patients with aggravating tumor and other serious consumptive disease, and who are subject to infection and bleeding.
* With serious protopathy or disease of cardiovascular, liver, renal, gastrointestinal, hematological systems and so on.
* Pregnant women or women in lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The proportion of participants reporting complete absence of dyspeptic symptoms | at 16 weeks after inclusion

SECONDARY OUTCOMES:
validated Leeds Dyspepsia Questionnaire | 4, 8, 16, 20, 24 weeks after inclusion
Nepean dyspepsia index | 4, 8, 16, 20, 24 weeks after inclusion
adverse events in each group | 4 weeks after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Fan-rong Liang, MD, Study Chair — Chengdu University of TCM
Locations (1):
- Chengdu University of TCM, Chengdu, Sichuan, China

REFERENCES:
- [Background] Ma TT, Yu SY, Li Y, Liang FR, Tian XP, Zheng H, Yan J, Sun GJ, Chang XR, Zhao L, Wu X, Zeng F. Randomised clinical trial: an assessment of acupuncture on specific meridian or specific acupoint vs. sham acupuncture for treating functional dyspepsia. Aliment Pharmacol Ther. 2012 Mar;35(5):552-61. doi: 10.1111/j.1365-2036.2011.04979.x. Epub 2012 Jan 16. PMID 22243034
- [Derived] Zheng H, Xu J, Li J, Li X, Zhao L, Chang X, Liu M, Gong B, Li X, Liang F. Acupuncture for patients with functional dyspepsia: study protocol of a randomised controlled trial. BMJ Open. 2013 Jul 30;3(7):e003377. doi: 10.1136/bmjopen-2013-003377. PMID 23901030